CLINICAL TRIAL: NCT00094146
Title: Sandostatin LAR® Depot in Patients With Primary Insulin Hypersecretion (PIH) and at Least Moderate Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSMS995GUS20; US20
Record Dates: First submitted 2004-10-14; First posted 2004-10-15 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2004-10

CONDITIONS: Primary Insulin Hypersecretion; Obesity
Keywords: Primary Insulin Hypersecretion; PIH; Obesity
MeSH Terms: conditions — Obesity | interventions — Octreotide

INTERVENTIONS:
Drug: Sandostatin LAR Depot

SUMMARY:
This study is in patients with at least moderate obesity (Body Mass Index [BMI] > 30 kg/m2 or approximately 30 or more pounds overweight) and who also produce too much insulin (insulin stores sugar as fat). Sandostatin LAR® Depot suppresses insulin, and is being developed to help with weight loss in people who find it hard to lose weight on their own because they produce too much insulin.

The main purpose of the study is to find the lowest dose of Sandostatin LAR® Depot that safely helps overweight people lose weight. The study will also compare weight loss in obese patients who receive one of three different dosages of Sandostatin LAR Depot or placebo.

ELIGIBILITY:
Inclusion Criteria:

You may qualify for this study if you:

* are between the ages of 18-70 (male or female)
* are at least moderately obese (BMI > 30 kg/m2 or approximately 30 or more pounds overweight)
* and pass an oral glucose tolerance test (a 3 hour test to determine if your body produces too much insulin)

Exclusion Criteria:

You are not qualified for this study if you:

* have diabetes
* have been able to lose weight with diet and exercise alone
* have previously received Sandostatin LAR® Depot

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2002-01; Study Completion 2002-12

PRIMARY OUTCOMES:
The percent change at baseline compared to 6 months in body weight

SECONDARY OUTCOMES:
Compare changes from baseline and at 6 months in body mass index (BMI), percentage of total body fat percentage of abdominal fat, leptin, and waist-to-hip ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hedrick, MBA, Study Director — Novartis
Locations (3):
- United States (3):
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - University of Tennessee, Memphis, Tennessee
  - University of Wisconsin Beers-Murphy Clinical Nutrition Clinic, Madison, Wisconsin

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=717